CLINICAL TRIAL: NCT00002074
Title: Multicenter Comparison of Fluconazole (UK-49,858) and Amphotericin B as Maintenance Treatment for the Prevention of Relapse of Cryptococcal Meningitis in Patients With Acquired Immunodeficiency Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012D; 056-157
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-05

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Fluconazole; Acquired Immunodeficiency Syndrome; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole; Amphotericin B

INTERVENTIONS:
Drug: Fluconazole
Drug: Amphotericin B

SUMMARY:
To compare the safety and effectiveness of fluconazole and amphotericin B as maintenance treatment for preventing the relapse of cryptococcal meningitis in patients with AIDS.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antivirals such as zidovudine.
* Prophylaxis (including aerosolized pentamidine) for Pneumocystis carinii pneumonia (PCP).
* Pfizer must be notified if the patient is receiving ganciclovir (DHPG) at entry.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Patients must be oriented to person, place, and time, and able to give written informed consent.

* Patients must have had an acute episode of cryptococcal meningitis that was documented by recovery and identification of Cryptococcus neoformans from lumbar cerebrospinal fluid (CSF) culture within 6 months prior to entry.
* Minimum total dose of 15 mg/kg of amphotericin B must have been given (either alone or in combination with flucytosine) during primary therapy.
* Patients need not be receiving amphotericin B at the time of randomization but must begin study maintenance therapy within 6 weeks of completion of primary amphotericin B therapy. Patients may receive maintenance amphotericin B during the period between completion of primary therapy and study entry.

Prior Medication:

Allowed:

* Antivirals such as zidovudine (AZT).
* Prophylaxis (including aerosolized pentamidine) for Pneumocystis carinii pneumonia (PCP).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Clinical evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease.

Concurrent Medication:

Excluded:

* Ketoconazole.
* Fluconazole.
* Itraconazole.
* Miconazole.
* Any systemic imidazole or azole for more than 7 days after initiation of primary therapy for cryptococcosis.
* Intrathecal amphotericin B.
* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Clinical evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease.
* Inability to take oral medications reliably.

Prior Medication:

Excluded:

* Ketoconazole.
* Fluconazole.
* Itraconazole.
* Miconazole.
* Any systemic imidazole or azole for more than 7 days after initiation of primary therapy for cryptococcosis.
* Intrathecal amphotericin B.
* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.
* Any exceptions to these prohibitions of concomitant medications must be approved by Pfizer Central Research.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (39):
- United States (38):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Tucson Veterans Administration Med Ctr, Tucson, Arizona
  - Dr Richard Meyer, Los Angeles, California
  - Davies Med Ctr, San Francisco, California
  - Dr Paul Rothman, Sherman Oaks, California
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Florida College of Medicine, Gainesville, Florida
  - Univ of South Florida, Tampa, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - DeKalb Gen Hosp, Decatur, Georgia
  - Shallowford Hosp, Decatur, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Dr Michael Bach, Portland, Maine
  - Univ of Maryland / Inst of Human Virology, Baltimore, Maryland
  - New England Med Ctr, Boston, Massachusetts
  - Univ Hosp, Boston, Massachusetts
  - Ann Arbor Veterans Administration Med Ctr, Ann Arbor, Michigan
  - Harper Hosp, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Saint Michael's Med Ctr, Newark, New Jersey
  - Albany Med College / AIDS Treatment Ctr, Albany, New York
  - Jewish Hosp Ctr Affiliation, Jamaica, New York
  - Cabrini Med Ctr, New York, New York
  - Chelsea Village Med Ctr, New York, New York
  - Columbia Univ, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bowman Gray School of Medicine / North Carolina Baptist Hosp, Winston-Salem, North Carolina
  - Cincinnati Veterans Adm Med Ctr / Univ Hosp, Cincinnati, Ohio
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas
  - United States Air Force Med Ctr, Lackland Air Force Base, Texas
  - Southwest Texas Methodist Hosp, San Antonio, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Richmond AIDS Consortium, Richmond, Virginia
  - CHG-118 Group Health / Cooperative of Puget Sound, Seattle, Washington
  - Dr Philip C Craven, Tacoma, Washington
- Saint Michael's Hosp, Toronto, Ontario, Canada

REFERENCES:
- [Background] Powderly WG, Saag MS, Cloud GA, Robinson P, Meyer RD, Jacobson JM, Graybill JR, Sugar AM, McAuliffe VJ, Follansbee SE, et al. A controlled trial of fluconazole or amphotericin B to prevent relapse of cryptococcal meningitis in patients with the acquired immunodeficiency syndrome. The NIAID AIDS Clinical Trials Group and Mycoses Study Group. N Engl J Med. 1992 Mar 19;326(12):793-8. doi: 10.1056/NEJM199203193261203. PMID 1538722
- [Background] Saag MS, Powderly WG, Cloud GA, Robinson P, Grieco MH, Sharkey PK, Thompson SE, Sugar AM, Tuazon CU, Fisher JF, et al. Comparison of amphotericin B with fluconazole in the treatment of acute AIDS-associated cryptococcal meningitis. The NIAID Mycoses Study Group and the AIDS Clinical Trials Group. N Engl J Med. 1992 Jan 9;326(2):83-9. doi: 10.1056/NEJM199201093260202. PMID 1727236